CLINICAL TRIAL: NCT04535505
Title: Establishment a Nucleic Acid Rapid Detection Technology Platform for Detecting Pathogenic Bordetella and Its Drug Resistance Genes
Brief Title: Pathogenic Bordetella Rapid Detection
Status: Withdrawn | Type: Observational
Why Stopped: Not as a lead unit
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: BRD1.0
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pertussis
Keywords: Pertussis；Children；Diagnostic test；CPA; CRISPR
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab of a suspected pertussis patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pertussis test population: People with clinical diagnosis of suspected pertussis in outpatient and ward in the Children's Hospital of Fudan University will be collected as study subjects. Their nasopharyngeal swabs will be collected. Bordetella isolation culture and identification method is the gold standard, and the new CPA platform based on CRISPR technology is the method to be tested. Diagnostic values of this research platform would be detected.
  Interventions: Diagnostic Test: Detection pathogenic pertussis by cross primer constant temperature amplification (CPA) and drug resistant genes of erythromycin by CRISPR technology

INTERVENTIONS:
Diagnostic Test: Detection pathogenic pertussis by cross primer constant temperature amplification (CPA) and drug resistant genes of erythromycin by CRISPR technology — This is an observational study and there are no interventions. The purpose of the study is to compare the accuracy （including sensitivity and specificity）of the new CPA platform based on CRISPR technology detection method and the gold standard in detecting pertussis patients.

SUMMARY:
A CPA platform based on the CRISPR technology is going to established to achieve the goal of detecting pathogenic bordetella and drug resistance genes in one step. The accuracy of this platform will be checked through prospective diagnostic test evaluation methods. Bordetella pertussis isolation culture and identification would be set as a gold standard method.

DETAILED DESCRIPTION:
Pertussis is an acute respiratory infectious disease caused by bordetella pertussis. Although it is a vaccine-preventable disease, outbreaks and epidemic cases of whooping cough worldwide have been reported from time to time. Bordella parapertussis, Bodella bronchiseptica, and bordetella hosei can cause pertussis-like diseases with symptoms similar to those of whooping cough. The clinical manifestations are difficult to distinguish, and they are easily reported as cases of whooping cough through the infectious disease network.

The diagnosis of the infectious diseases caused by the four pathogenic bodella mainly relies on laboratory pathogenic testing. At present, the laboratory tests of bordetella that can be carried out in the clinical microbiology laboratory include culture, bordetella pertussis specific antibody (PT-IgG) serological detection, and bordetella pertussis nucleic acid PCR detection. However, none of them meet the requirements of early diagnosis.

Cross primer constant temperature amplification (CPA) is nucleic acid constant temperature amplification technology with independent property rights. The fully automated nucleic acid detection platform equipped with CPA technology would make the detection of four pathogenic bordetella easy, quick and safe and accurate.

As pathogenic bodella is difficult to cultivate and there is no standard for drug susceptibility test. Studies have shown that 57.4% of the isolated clinical isolates of bordetella pertussis have MIC value for erthomycin ≥256 μg/mL , and 23s rRNA 2047 site adenine (A) were mutated to guanine (G).CRISPR/Cas is an immune system in bacteria that can specifically recognize invading nucleic acids and shear them. The CRISPR technology developed based on the CRISPR/Cas principle can detect single point mutations in genes.

The hypothesis that 4 pathogenic bordetella and their erythromycin resistance would be detected in one testing platform simultaneously. The accuracy, reliability, predictive value of this platform would be checked through prospective diagnostic test evaluation methods. Bordetella pertussis isolation culture and identification would be as the gold standard method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with continuous cough (paroxysmal cough) for more than 1 week, peripheral white blood cell 18×109/L (infants and young children), or> 15×109/L (children), ineffective use of cephalosporin antibacterial drugs，and these patients whose nasopharyngeal swabs are collected for routine bordetella culture identification and drug susceptibility testing would be included as research object.

Exclusion Criteria:

* Patients with pertussis are suspected clinically but no nasopharyngeal swab specimens are collected or patients with pertussis are clinically excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 600 cases of suspected pertussis clinically diagnosed in the outpatient clinic and ward of Children's Hospital of Fudan University would be enrolled. The enrollment would start in October 2021 and end in June 2022. Patients who are admitted to the Children's Hospital of Fudan University during the enrollment period and are clinically suspected of pertussis would be the research objects. There are no special requirements for gender of the enrolled patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the new CPA platform based on CRISPR technology, including sensitivity and specificity | At enrollment
  Bordetella pertussis isolation culture and identification would be taken as gold standard. The enrolled subjects would receive the detection of this research platform detection method and the gold standard at the same time. The measurement indexes are sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanqing Wang, Phd, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No